CLINICAL TRIAL: NCT02297425
Title: Phase 1/2 Open Label Study Of Pf 06459988 (Epidermal Growth Factor Receptor T790m Inhibitor) In Patients With Advanced Epidermal Growth Factor Receptor Mutant (Del 19 Or L858r + - T790m) Non Small Cell Lung Cancer
Brief Title: A Study For Patients With EGFRm (Epidermal Growth Factor Receptor Mutant) Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7711001; T790M (Other: Alias Study Number)
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Advanced EGFRm (Del 19 or L858R +/- T790M) NSCLC
Keywords: NSCLC, Non-Small Cell Lung Cancer, EGFRm, Epidermal Grown Factor Receptor mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — PF-06459988

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single agent - study drug (Experimental): The study will evaluate single-agent PF-06459988
  Interventions: Drug: PF-06459988

INTERVENTIONS:
Drug: PF-06459988 — The study will evaluate PF-06459988 PO (tablets) continuous daily dosing in 21 day cycles. The starting dose for PF-06459988 will be 50 mg PO daily. The escalation/de-escalation rules will follow the modified toxicity probability interval method with adjustments using the DLT rate and maximum size per dose level of 10 patients

SUMMARY:
Phase 1 - open label, multi-center, non-randomized, safety, pharmacokinetic and pharmacodynamics dose escalation study of PF-06459988 as a single agent in patients with advance EGFRm NSCLC (del 19, L858R, +/- T790M). The resulting PF-06459988 dose selected from the phase 1 portion will undergo a series of sub-studies to fully characterize the impact of food, antacid and CYP3A4 inhibitors/inducers. The PK studies are in addition to the MTD expansion and will be completed prior to the initiation of Phase 2. Phase 2 is an open label, multi-center single-arm study of PF-06459988 for the assessment of antitumor activity in patients with advanced EGFRm (del 19 or L858R) NSCLC with T790M.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of histological or cytologically confirmed diagnosis of locally advanced or metastatic EGFRm (del19 or L858R) NSCLC that is resistant to standard therapy. Patients must have progressed on treatment with an EGFR TKI, and may have also received other line of therapy.
* Tissue available (formalin fixed paraffin embedded (FFPE) block or 10 unstained sections (5 micron)
* Patients must be willing to participate in additional PK studies as required (cohort dependent); patients will be informed of which PK studies are required prior to consenting for study participation
* Adequate Bone Marrow Function (Complete Blood Count laboratory test results)
* Adequate Liver Function (Laboratory test)

Exclusion Criteria:

* Previously diagnosed brain metastases, unless the patient has completed their treatment and has recovered from the acute effects of radiation therapy or surgery prior to the study registration, have discontinued corticosteroid treatment for these metastases for at least 2 weeks and are neurologically stable
* Systemic anti-cancer therapy within 4 weeks of starting study treatment excluding EGFR TKIs. Patients on EGFR TKIs must discontinue the agent for a minimum of 5 days prior to starting study drug
* Hypertension that cannot be controlled by medication (150/100 mmHg despite optimal medical therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose-limiting toxicities (DLT) (phase 1) | up to 21 days
  The target probability of DLT at MTD will be 30%
Number of Participants With Objective Response (phase 2) | Time from first dose of study drug to objective response of CR or PR up to 24 months
  Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. PR are those as noted in the RECIST Criteria: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions

SECONDARY OUTCOMES:
Number of Participants With Objective Response for those patients with measurable disease (phase 1) | time from first dose of study drug until objective response of CR or PR up to 24 months
  Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. PR are those PR are those as noted in the RECIST Criteria: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions
Progression-Free Survival (PFS) - Phase 2 | time from first dose of study drug until Disease Progression or death (whichever first) up to 24 months
  The period from study entry until disease progression, death or date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7711001&StudyName=A%20Study%20For%20Patients%20With%20EGFRm%20%28Epidermal%20Growth%20Factor%20Receptor%20Mutant%29%20Lung%20Cancer